CLINICAL TRIAL: NCT05784207
Title: An In Silico Trial to Evaluate Prospectively the Performance of a Radiomics Algorithm for UIP Compared to Medical Doctors
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: ISTRU
Record Dates: First submitted 2021-05-19; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease; Radiomics
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IPF/UIP_CT based: patients with an ILD and a pathological UIP pattern and a final diagnosis of IPF
  Interventions: Other: Radiomics model to classify between IPF with UIP pattern and ILDs without UIP pattern
- IPF/UIP_Biopsy based: patients with a final diagnosis of IPF but a less typical HRCT pattern( lung biopsy required for the diagnosis)
  Interventions: Other: Radiomics model to classify between IPF with UIP pattern and ILDs without UIP pattern
- ILD but not IPF and prove by biopsy not UIP: patients with an ILD and a pathological non-UIP pattern
  Interventions: Other: Radiomics model to classify between IPF with UIP pattern and ILDs without UIP pattern
- Normal: Normal healthy patients
  Interventions: Other: Radiomics model to classify between IPF with UIP pattern and ILDs without UIP pattern

INTERVENTIONS:
Other: Radiomics model to classify between IPF with UIP pattern and ILDs without UIP pattern — The aim is to evaluate the performance of AI with the performance of doctors

SUMMARY:
The purpose of this study is to compare AI performance to doctor's performance in the evaluation of IPF/UIP and ILDs without UIP(proven by biopsy).

ELIGIBILITY:
Inclusion Criteria:

- the availability of non-contrast-enhanced HRCT

Exclusion Criteria:

* the use of contrast enhancement
* images containing metal or motion artifacts
* Images reconstructed with a slice thickness larger than 1.5 mm

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had HRCT and shown IPF/UIP in CT images, or patients who is suspected to have IPF based on MMD and proved by lung biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The performance of Radiomics algorithm compared to the ground truth | May 2021
  Reporting the performance measure: accuracy

SECONDARY OUTCOMES:
Comparing the performance of the radiomics algorithm to that of physicians | June 2021
  Correctness of the diagnosis - the most probable thin-section pattern (dichotomous outcome: yes or no)

OTHER OUTCOMES:
Comparing the performance of radiomics algorithm to that of individual doctor | June 2021
  Correctness of the diagnosis - the most probable thin-section pattern (dichotomous outcome: yes or no)
Comparing the reproducibility of diagnosis between the doctors | June 2021
  Measuring the concordance in diagnosis in between the physicians, and for each physician separately, using the Concordance correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands